CLINICAL TRIAL: NCT04163393
Title: R-One Efficiency For PCI Evolution With Robotic Assistance
Acronym: R-EVOLUTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robocath (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROB-01
Record Dates: First submitted 2019-10-15; First posted 2019-11-14 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-One (Experimental): Patients treated with robotic assistance
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: Percutaneous Coronary Intervention using R-One assistance

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — PCI with robotic assistance
Device: Percutaneous Coronary Intervention using R-One assistance — PCI with robotic assistance

SUMMARY:
This study is a Prospective, Multi-center, Single-arm clinical study, in patients with Coronary Artery Disease, including patients with silent ischemia (excluding STEMI), who qualify for elective Percutaneous Coronary Intervention (PCI), aimed to assess the Safety and Efficacy of the R-One device in elective PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Candidate for PCI;
* Presence of a de novo coronary artery stenosis of ≥ 50% and <100% in a native coronary artery indicated and suitable for stent implantation;
* The vessel has a reference vessel diameter ranging from 2.5 mm to 4.0 mm;
* The target lesion length allows for treatment with a single stent up to 38 mm in length;
* Up to 2 target vessels each with a single target lesion requiring a single stent per lesion and treatable within a single procedure may be included (no further staged procedure allowed);
* The patient provides written informed consent as approved by the applicable Ethics Committee and is willing to comply with all study requirements including 30 days follow-up.

Exclusion Criteria:

* Target lesion has TIMI flow < 3;
* Treatment of in-stent restenosis, or prior stent in the target vessel proximal to the target lesion;
* More than one target lesion per vessel requiring treatment at the time of procedure;
* Target lesion is a bifurcation requiring balloon or stent implantation of the side branch, with a side-branch RVD of ≥1.5 mm with a DS ≥50% at or within 5 mm its origin, or RVD ≥2.0 mm regardless of the presence of side branch disease;
* Target lesion is located in left main coronary artery, or any left main stenosis > 30%;
* Target lesion is within 5 mm of the ostial LAD, ostial LCX or ostial RCA;
* Severe vessel tortuosity;
* Severe vessel calcification;
* STEMI, cardiopulmonary resuscitation or cardiogenic shock within 48 hours of the procedure;
* Presence of visible thrombus;
* Need for any procedure other than balloon angioplasty or stenting (e.g. atherectomy, laser, are excluded);
* Patients under judicial protection, tutorship or curatorship (for France only);
* Any patient participating in another clinical study evaluating a drug or a medical device (except registries for which the primary endpoint has not been evaluated;
* Pregnant and breast-feeding women or intention to become pregnant prior to completion of all follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint: Number of patients with absence of Intra-procedural complications (Dissection, Thrombus, Air embolus, traumatic aorta) | Peri-procedure
  Absence of Intra-procedural complications (Dissection >/= NHLBI type D, perforation, decrease of TIMI flow (</= 2), acute occlusion, visible thrombus formation, significant air embolus, traumatic aortic or Left Main dissection by guiding catheter
Efficacy Endpoint: Number of Patients with Procedure technical success | During Procedure
  Procedure technical success defined as the successful advancement and retraction of all PCI devices (guidewires, balloon catheters and stents) and the successful treatment of all the target lesions using the R-One system and without conversion to manual operation

SECONDARY OUTCOMES:
Number of patients with Absence of each type of Intra-procedural complication (Dissection, Thrombus, Air embolus, traumatic aorta) | During Procedure
  Component of the Primary Safety Endpoint: Absence of Intra-procedural complications (Dissection >/= NHLBI type D, perforation, decrease of TIMI flow (</= 2), acute occlusion, visible thrombus formation, significant air embolus, traumatic aortic or Left Main dissection by guiding catheter
Procedure duration | During Procedure
  Time between arterial sheath introduction and sheath removal
Robot duration | During Procedure
  From the time when the robot begins to manipulate the guidewire to the time when the last guidewire is removed
Radiation exposure using dosimeters (Patient Radiation, Robot Dose, Procedure Dose) | During Procedure
  Patient and Operator
Contrast Volume in mL | During Procedure
  Measure of the volume of injected contrast media
Rate of Bleeding or Vascular Complications | Up to 1 month
  BARC definition
Rate of Device Oriented Composite Criteria (Cardiovascular Death, Myocardial Infarction (peri-procedural and spontaneous), non clearly attributed to a non target or clinically driven target lesion revascularization) | Post-Procedure, 1 month
  ARC 2 definition: Cardiovascular Death, Myocardial Infarction (peri-procedural and spontaneous), non clearly attributed to a non target or clinically driven target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (6):
- Het Ziekenhuisnetwerk Antwerpen vzw, Antwerp, Belgium
- France (3):
  - CHU Caen Normandie, Caen
  - CHU Rouen, Rouen
  - Clinique Pasteur, Toulouse
- INCCI, Luxembourg, Luxembourg
- Maastad Ziekenhuis, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durand E, Sabatier R, Smits PC, Verheye S, Pereira B, Fajadet J. Evaluation of the R-One robotic system for percutaneous coronary intervention: the R-EVOLUTION study. EuroIntervention. 2023 Apr 3;18(16):e1339-e1347. doi: 10.4244/EIJ-D-22-00642. PMID 36602883